CLINICAL TRIAL: NCT03659409
Title: Investigating the Impact of Mindfulness on the Physiological and Psychological Well-being of Stroke Survivors and Their Caregivers.
Brief Title: Stroke Of Mindfulness: Investigating Physiological and Psychological Well-being
Acronym: SOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016/2361
Record Dates: First submitted 2018-05-13; First posted 2018-09-06 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Stress; Anxiety; Depression
Keywords: Mindfulness; Stroke Survivors; Caregivers
MeSH Terms: conditions — Stroke; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive either the intervention or treatment as usual. The intervention is for 4 weeks, and 3 months from the start of the intervention, participants who were assigned to the treatment as usual group will receive the same intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Intervention (Experimental): 4 weekly 2-hour sessions. Participants will be introduced, taught and guided in practice of mindfulness-based interventions that are focused on their (1) breath, (2) senses, (3) body and bodily movements, (4) feelings of empathy and compassion.
  Interventions: Behavioral: Mindfulness-Based Intervention
- Treatment Waitlist Group (Other): Participants will receive no intervention, except for a baseline follow-up at the start and again at the end of the first phase. 2 months after the end of the first intervention phase, participants in this group will receive the same mindfulness-based intervention for 4 weeks.
  Interventions: Behavioral: Waitlist - Mindfulness-Based Intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — 4 weekly 2-hour sessions. Participants will be introduced, taught and guided in practice of mindfulness-based interventions that are focused on their (1) breath, (2) senses, (3) body and bodily movements, (4) feelings of empathy and compassion.
  Arms: Mindfulness Based Intervention
Behavioral: Waitlist - Mindfulness-Based Intervention — Participants in this group will only receive the Mindfulness-Based Intervention 3-months after they have started the study and baseline measurements. While participants in the Intervention Arm are receiving the treatment, this group will receive No intervention for the first four weeks and will continue as treatment as usual until it is their turn to receive the Intervention.
  Arms: Treatment Waitlist Group

SUMMARY:
This study evaluates the impact of mindfulness-based interventions on psycho-social and physiological well-being among stroke survivors and their family caregivers. This study will employ a treatment wait-list cross-over design, with half the participants randomized to receive the intervention first (treatment group), while the other half receives the interventions 2 months following the end of the treatment phase (wait-list group).

DETAILED DESCRIPTION:
Stroke survivors face many concerns, including the physical, psychological, cognitive and psychosocial consequences of stroke, as well as impaired function and quality of life. Also important for stroke survivors is the possibility of recurrence that may result in death and further disability. Survivors depend on their caregivers to provide assistance for daily living tasks, emotional support and taking on new roles and responsibilities with changing social dynamics, often causing long-term strain.

Mindfulness-based interventions (MBIs) are psychotherapeutic interventions which have been shown to improve psychological, physiological and psychosocial outcomes such as anxiety, depression, mental fatigue, blood pressure and overall quality of life. However, data is limited for stroke survivors and their caregivers, especially in Asians. This study will evaluate the impact of MBIs on the psychological well-being and perceived quality of life among stroke survivors and their family caregivers in Singapore.

This study employs a randomized treatment-waitlist crossover design with outcome measures administered before and after the intervention as well as at 3 months follow-up for the treatment group.

The intervention consists of 4 weekly 2-hour mindfulness sessions. Participants will be introduced, taught and guided in practice of mindfulness-based interventions that are focused on their (1) breath, (2) senses, (3) body and bodily movement, (4) feelings of empathy and compassion. Pre- and post-intervention questionnaires will be conducted to assess symptoms associated with depression, anxiety, stress and perceived quality of life. Blood pressure and heart rate variability recordings before and after intervention will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Stroke Survivors
* Family Caregivers
* Able to speak and understand English Fluently
* Comprehends and provides consent independently

Exclusion Criteria:

* Cognitively impaired individuals with a MMSE Score of less than 20, MoCA score of less than 23
* Depression and Anxiety Stress Scale Scores, DASS, Depression >7, Anxiety >8, and Stress >13

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Cohen Perceived Stress Scale | Past 1 Month
  A 10-item measure evaluating the perception of stress.
Centre for Epidemiologic Studies Depression Scale (CES-D) | Past 1 Week
  A 20-item measure for epidemiological research on depression.
Stroke Specific Quality of Life Scale (SS-QOL) | Past 1 Month
  A 49-item self-report questionnaire designed to measure the heath related quality of life specific to stroke survivors across 12 domains.
Stroke Impact Scale (SIS) | 1 week
  A 64-item questionnaire that assesses across 8 domains
Short-Form-36 (SF-36) | A range from the past 4 to 52 weeks
  A 36-item self-report survey of health, including physical and mental health. Higher scaled scores reflect better quality of health.

SECONDARY OUTCOMES:
Zarit Burden Interview | Past 1 Month
  A 22-item self-report questionnaire to measure for level of caregiver burden or stress.
Five Facet Mindfulness Questionnaire | Past 1 Month
  This 39-item instrument is based on a factor analytic study of five independently developed mindfulness questionnaires. The analysis yielded five factors that appear to represent elements of mindfulness as it is currently conceptualized. The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
Big Five Personality Inventory | Past 1 Month
  44-item inventory that measures an individual on the Big Five Factors (dimensions) of personality (Goldberg, 1993). Each of the factors is then further divided into personality facets.

OTHER OUTCOMES:
Mental Fatigue Scale (MFS) | 1 Month
  A 15-item questionnaire that cover the most common symptoms that occur after brain injury such as that sustained after a stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Kinjal Doshi, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Preliminary data to inform design of future studies.